CLINICAL TRIAL: NCT07256223
Title: A Single-Arm, Multicenter, Prospective Clinical Study of Envafolimab Combined With Lenvatinib as First-Line Therapy in Renal Cell Carcinoma Patients With Liver Metastases
Brief Title: A Clinical Trial of Envafolimab Combined With Lenvatinib for Kidney Cancer With Liver Spread
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huadong Hospital (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Director of Urology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-RCC-001
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Clear Cell Renal Cell Cancer (ccRCC); Liver Metastasis
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab+Lenvatinib (Experimental): Envafolimab+Lenvatinib
  Interventions: Drug: Envafolimab+Lenvatinib

INTERVENTIONS:
Drug: Envafolimab+Lenvatinib — To evaluate the efficacy and safety of envafolimab in combination with lenvatinib for the treatment of patients with clear cell renal cell carcinoma (ccRCC) accompanied by liver metastases.

SUMMARY:
This is an open-label, single-arm, prospective, multicenter clinical study designed to evaluate the efficacy and safety of envafolimab in combination with lenvatinib for the treatment of patients with clear cell renal cell carcinoma (ccRCC) accompanied by liver metastases. The Department of Urology at Fudan University Shanghai Cancer Center serves as the primary research center.

DETAILED DESCRIPTION:
The study procedure comprises three phases: a screening period, a treatment period, and a follow-up period. Patients with previously untreated advanced clear cell renal cell carcinoma and liver metastases will be screened. Those who meet the inclusion criteria and provide written informed consent will receive treatment. The treatment regimen consists of envafolimab combined with lenvatinib administered over 8 treatment cycles, with each cycle defined as 14 days. enrolled patients will undergo biopsy of liver metastases before the first dose and after 8 cycles of treatment (or upon confirmation of disease progression). Imaging examinations of the kidneys and liver will be conducted during the screening period, after 4 cycles of treatment, and after 8 cycles of treatment. Following the initiation of therapy, systemic imaging will be performed every 6 months. Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. Safety evaluations will be based on the Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, with relevant laboratory tests performed during each treatment cycle. Adverse events will be recorded from the time of enrollment until 30 days after the last dose. For serious adverse events or those considered related to envafolimab, the recording period will be extended to 90 days after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for enrollment in the study:

Provide written informed consent prior to any study-specific procedures.

Aged between 18 and 75 years, inclusive.

Histologically confirmed clear cell renal cell carcinoma with radiologically documented liver metastases, and having received no prior systemic antitumor therapy.

Presence of at least one measurable liver metastasis lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (with the longest diameter ≥ 10 mm on computed tomography scan for non-lymph node lesions).

Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Life expectancy of ≥ 3 months.

Voluntarily agree to participate in the study with good compliance.

Adequate organ and bone marrow function, defined as follows:

Hematological:Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count (PLT) ≥ 70 × 10⁹/L; Hemoglobin (HGB) ≥ 90 g/L.

Hepatic:Serum total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN; Serum albumin ≥ 28 g/L; Alkaline phosphatase (ALP) ≤ 5 × ULN. (Subjects who meet the above criteria after conventional liver-protecting therapy and remain stable for at least one week, as assessed by the investigator, may be enrolled.)

Renal:Serum creatinine (Cr) ≤ 1.5 × ULN, or calculated creatinine clearance ≥ 50 mL/min (using the standard Cockcroft-Gault formula).

Coagulation:International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN, and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. (For subjects receiving anticoagulant therapy, enrollment is permitted if the PT and INR are within the therapeutic range intended by the anticoagulant medication.)

Exclusion Criteria:

History of or concurrent other malignancies, except for appropriately treated carcinoma in situ or non-melanoma skin cancer with evidence of cure.

Prior systemic antitumor therapy for advanced disease (including antiangiogenic agents and immunotherapy), with the exception of palliative radiotherapy or preoperative PD-1 neoadjuvant therapy.

Presence of metastatic lesions meeting any of the following: unifocal organ metastasis numbering more than 3, or total systemic metastatic foci exceeding 5.

Known history of hypersensitivity to any component of the investigational drug products.

Poorly controlled cardiac symptoms or diseases, including: (1) heart failure of New York Heart Association (NYHA) Class II or higher; (2) unstable angina pectoris; (3) myocardial infarction within the past year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.

Active infection, or unexplained fever > 38.5°C occurring during the screening period or before the first dose (subjects with fever determined by the investigator to be tumor-related may be enrolled).

Administration of live vaccines within 4 weeks prior to the first dose of study treatment or anticipated during the study period.

History of substance abuse, drug addiction, or chronic alcohol abuse.

Any condition that, in the judgment of the investigator, would preclude participation in the study. This includes severe concomitant conditions (including psychiatric disorders) requiring treatment, significant laboratory abnormalities, or social/familial factors that could compromise subject safety or adherence to protocol requirements, including data and sample collection

.

Active hepatitis B infection.

Active systemic autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
ORR of liver lesions | 2 years
  Objective Response Rate (ORR) of liver lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
DCR of liver lesions | 2 years
  DCR of liver lesions
Progression-Free Survival (PFS) | 2 years
  Progression-Free Survival (PFS)
1-year Overall Survival (OS) rate | 2 years
  1-year Overall Survival (OS) rate